CLINICAL TRIAL: NCT03929887
Title: Multicenter Prospective Cohort of Kidney Biopsy for Glomerular Disease Research
Brief Title: KOrea Renal Biobank NEtwoRk System TOward NExt-generation Analysis
Acronym: KORNERSTONE
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); KangWon National University Hospital (Other); Keimyung University Dongsan Medical Center (Other); SMG-SNU Boramae Medical Center (Other); Seoul National University Bundang Hospital (Other); Severance Hospital (Other); Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Dong Ki Kim, Professor, Seoul National University Hospital
Other Study IDs: KORNERSTONE
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Glomerular Disease; Minimal Change Disease; IgA Nephropathy; Membranous Nephropathy; Focal Segmental Glomerulosclerosis; Lupus Nephritis; Crescentic Glomerulonephritis
Keywords: Glomerular disease; sample repository; clinical data; digital pathology repository; web-based database
MeSH Terms: conditions — Nephrosis, Lipoid; Glomerulonephritis, IGA; Glomerulonephritis, Membranous; Glomerulosclerosis, Focal Segmental; Lupus Nephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — plasma, serum, genomic DNA, buffy coat, urine, stool, glomerular cDNA, tubulointerstitial cDNA, kidney biopsy slides (digitalized)
  These sample are acquired at kidney biopsy, annually afterwords, and at the time of clinical endpoint if possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- KORNERSTONE: Glomerulonephritis (GN) such as Minimal change disease (MCD), focal segmental glomerulosclerosis (FSGS), Membranous nephropathy (MN), and Immunoglobulin A nephropathy (IgAN)
  Participants enrolled in KORNERSTONE with a biopsy proven GN.
  Eligible participants must be scheduled for a clinically indicated renal biopsy.
  Interventions: Other: Kidney Biopsy

INTERVENTIONS:
Other: Kidney Biopsy — Patients scheduled to undergo a clinically indicated kidney biopsy will be requested to consent to an additional renal core and various patient-derived samples.

SUMMARY:
Glomerulonephritis (GN) generates an enormous individual and social economic burden. However, the therapeutic options are largely based on clinical and pathological parameters and the individual response to therapy or prognosis is uncertain.

Recently, along with advances in molecular analysis and computational bioinformatics, genomic data from human renal biopsies could provide a strong foundation for the future of precision medicine in nephrology.

In response to a request for applications by the Ministry of Health and Welfare of Korea for the creation of Clinical Research Registry, multi-center N network has been established for prospective cohort with kidney biopsy samples (KORNERSTONE).

Through this Network the investigators hope to understand the fundamental biology of glomerulonephritis and aim to bank long-term observational data and corresponding biological data including genomic data from kidney tissues, and kidney pathologic data which is digitalized This database is archived to a web-based platform to access easily and further enrich for researchers.

DETAILED DESCRIPTION:
Glomerulonephritis (GN) such as Minimal change disease (MCD), focal segmental glomerulosclerosis (FSGS), Membranous nephropathy (MN), and Immunoglobulin A nephropathy (IgAN) has quite a common clinical presentation often results in renal insufficiency which generates an enormous individual and social economic burden.

However, the therapeutic options are largely based on clinical and pathological parameters and the individual response to therapy or prognosis is uncertain.

Recently, along with advances in molecular analysis and computational bioinformatics, genomic data from human renal biopsies could provide a strong foundation for the future of precision medicine in nephrology.

In response to a request for applications by the Ministry of Health and Welfare of Korea for the creation of Clinical Research Registry, a number of universities joined together to establish Korean Kidney Biopsy Network (KORNERSTONE).

Through this Network the investigators hope to understand the fundamental biology of glomerulonephritis and aim to bank long-term observational data and corresponding biological data including genomic data from kidney tissues, and kidney pathologic data which is digitalized This database is archived to a web-based platform to access easily and further enrich for researchers.

============ <Patient clinical data will be collected as follows>

1. Blood tests: CBC, Chemistry (Ca, P, Glucose, Total protein, Albumin, Uric acid), Electrolyte, Renal function (BUN, Creatinine, eGFR), Liver function (AST, ALT)
2. Immunologic blood tests: Complement 3, Complement 4, ASO, RF, Cryoglobulin, dsDNA, ANA
3. Urine tests: Urinalysis, Urine protein, Urine albumin, Urine creatinine
4. Radiologic tests: Kidney USG, Abdominal-pelvis computed tomography
5. Pathologic results
6. Treatment informations: treatment status, drug type, treatment duration
7. Quality of life questionnaire: Kidney Disease and Quality of Life Short Form survey (adults), PedsQL 4.0 Generic Core Scales (pediatrics)
8. Dietary questionnaire

ELIGIBILITY:
1. Inclusion criteria

   * Patient suspected of glomerular disease who received kidney biopsy in participating university medical centers
   * Children (age<18 years) also included
2. Exclusion criteria - Patients who previously received a kidney transplant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suspected of glomerular diseases who received kidney biopsy in participating university medical centres are eligible for inclusion in the KORNERSTONE.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | 60 months
  Documentation of death from any cause
Deterioration of renal outcomes | 60 months
  1. Doubling of serum creatinine compared to baseline serum creatinine
  2. 30% decline in follow-up estimated GFR (using the MDRD equation and/or the CKD-EPI equation) compared to baseline measurement
  3. End stage renal disease defined as estimated GFR ≤10cc/min, initiation of maintenance dialysis or kidney transplantation.
Improvement of clinical outcomes | 60 months
  Remission of glomerulonephritis and proteinuria <0.3g/day (pateint who have proteinuria<0.3g/day at baseline have no improvement in clinical outcomes)

SECONDARY OUTCOMES:
Malignancies | 60 months
  Any cancer diagnosis of the skin, hematopoietic system, or solid organ after enrollment
Infections, Serious and Systemic | 60 months
  Documented infection of any vital organ requiring the use of parenteral and/or oral antibiotics.
Acute Kidney Injury | 60 months
  Documented diagnosis of acute kidney injury as defined by the RIFLE criteria and/or renal failure requiring renal replacement therapy <3 months.
Hospitalization | 60 months
  Documented hospital admission, including observation for ≥24 hours.
Emergency Department/ Observation Unit Visit | 60 months
  Documented visit to an emergency department or observation unit that does not lead to hospitalization and is less than 24 hours.
Cardiovascular/Cerebrovascular event | 60 months
  Myocardial infarction; Congestive heart failure; Primary intractable serious arrhythmia; Peripheral vascular disease; Ischemic cerebrovascular accident; Hemorrhagic cerebrovascular accident; Thromboembolic event
New Onset Diabetes | 60 months
  Diagnosis of diabetes as indicated by 1 or more of the following not present at enrollment
  1. Documented diagnosis of diabetes in medical record
  2. Casual (non-fasting) blood glucose > 200 mg/dL c) Fasting blood glucose > 126 mg/dL d) 2 hour glucose > 200 after oral glucose tolerance test e) chronic use (>6 mos) hypoglycemic therapy outside of pregnancy f) Hemogloblin A1C >= 6.5%

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ki Kim, MD, PhD, Study Director — Seoul National University Hospital
Locations (6):
- South Korea (6):
  - KangWon National University Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Chung-Ang University Hosptial, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Kang E, Kim Y, Kim YC, Kim E, Lee N, Kim Y, Lee S, Han S, Choe M, Hwang JH, Lee S, Park JI, Park JT, Lim BJ, Lee JP, An JN, Ryu DR, Kim JH, Kang HG, Lee HS, Moon KC, Joo KW, Oh KH, Han SS, Lee H, Kim DK; KORNERSTONE Study Group. Biobanking for glomerular diseases: a study design and protocol for KOrea Renal biobank NEtwoRk System TOward NExt-generation analysis (KORNERSTONE). BMC Nephrol. 2020 Aug 26;21(1):367. doi: 10.1186/s12882-020-02016-z. PMID 32842999